CLINICAL TRIAL: NCT02230774
Title: Hydration Amongst Nurses and Doctors Oncall
Acronym: HANDsOn
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: European Hydration Institute (Other); Loughborough University (Other)
Responsible Party: Sponsor
Other Study IDs: 12118
Record Dates: First submitted 2014-07-14; First posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Dehydration
Keywords: hydration; cognitive function; doctors; nurses; Nurses and Doctors oncall
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and urine sampling
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- medical staff: Nurses and doctors oncall

SUMMARY:
The main purpose of this study is to assess and compare the hydration status of medical and nursing staff and to investigate the relationship between the hydration status, cognitive function and serum cortisol (marker of stress).

We hypothesise that a significant proportion of doctors and nurses will be dehydrated at the end of their working day. Some, as in other occupations, may be dehydrated at the start of their working day. This is likely to be associated with impairment in cognitive performance at the end of the working day compared to the beginning and expected to be more pronounced after a night shift. There may be less noticeable difference amongst nursing staff given the protected break time. Dehydration and associated impairment in cognition is of important clinical value as it can impact patient care. participants will be involved in the study for two shifts (one day and one night), aiming at 15 medical and 15 surgical nurses as well as 15 medical (total 15 day and 15 night shifts from each group) and surgical doctors (total 15 day and 15 night shifts from each group). Those that do not work both day and night shifts will participate for only one shift and a new participant will be recruited until target number of shifts is achieved.

DETAILED DESCRIPTION:
End points

1. To assess the hydration status of hospital staff nurses and doctors oncall at work by measuring the following:

   1. Urine and serum osmolality
   2. Urine mass produced during the shift
   3. Kidney function (U &Es)
   4. Bioimpedance measures

      2- To assess the effect of hydration on status of cognitive function and subjective feelings.

      3- To assess the association between hydration status on stress hormone (cortisol) levels.

      Inclusion criteria All medical and nursing staff working on acute medical and surgical admissions at the Queens Medical Centre Nottingham.

      Exclusion Criteria:

      Pregnancy Pre-existing kidney disease Patients on diuretics Unwell in the past 6 week with acute illness that warrants hospital admission or prescribed medication.

ELIGIBILITY:
Inclusion Criteria:

* All medical and nursing staff working on acute medical and surgical admissions at the Queens Medical Centre Nottingham

Exclusion Criteria:

* Pregnancy Pre-existing kidney disease Patients on diuretics Unwell in the past 6 week with acute illness that warrants hospital admission or prescribed medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurses and doctors oncall working on acute medical and surgical admissions wards at the Queens Medical Centre Nottingham
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Assess the prevalence of dehydration in nurses and doctors oncall. | Participants will be followed up for the duration of their shift, approximately 12- 14 hours.
  Using urine osmolality as a marker of hydration we aim to assess the prevalence of dehydration in health care professionals before and after day and night shifts. Comparing nurses and doctors oncall, day and night as well diffrence between those working in medical and surgical admissions.

SECONDARY OUTCOMES:
Impact of hydration status on cognitive function | Participants will be followed up for the duration of their shift, approximately 12- 14 hours.
  We aim to assess the impact of hydration on key executive cognitive before and after day and night shifts, comparing day and night using the following tests:
  * Visual search
  * Stroop
  * Sternberg
  * Corsi
The impact of hydration status on serum cortisol concentrations | Participants will be followed up for the duration of their shift, approximately 12- 14 hours.
  The impact of hydration status on serum cortisol concentrations as a surrogate marker of stress will be assessed before and after day and night shifts. with day and night shifts assessed separately given the diurnal variations in cortisol.

CONTACTS AND LOCATIONS:
Overall Officials: Dileep N Lobo, MBBS,DM,FRCS, Study Chair — University of Nottingham; Dileep N Lobo, MBBS,DM,FRCS, Principal Investigator — University of Nottingham
Locations (1):
- Queens Medical Centre, Nottingham, Nottinghamshire, United Kingdom